CLINICAL TRIAL: NCT03085446
Title: Two-armed, Single-blind Randomized Clinical Trial for Older Adults With Insomnia
Brief Title: Insomnia in Older Adults: Impact of Personalized, Diet-Induced Alterations in the Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: The Max Stern Academic College Of Emek Yezreel (Other); Migal, Galilee Technology Center (Other); Tel Hai College (Other); Clalit Health Services (Other); Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSHaifa
Record Dates: First submitted 2017-03-19; First posted 2017-03-21 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Health

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDM nutritional intervention (Experimental)
  Interventions: Behavioral: PDM nutritional intervention
- control (Experimental): General information on nutrition and health
  Interventions: Behavioral: General information on nutrition and health

INTERVENTIONS:
Behavioral: PDM nutritional intervention — personalized, diet-induced alterations in microbiota (PDM) for six months. (1) A 14-day running-in, no-treatment baseline assessment of all outcomes (T0); (2) A 6-month intervention period, with repeated assessments of all outcomes during the last two weeks of months 3 (T1) and 6 (T2). (3) A 12 month follow up (T3).
  Arms: PDM nutritional intervention
Behavioral: General information on nutrition and health — General information on nutrition and health for six months: (1) A 14-day running-in, no-treatment baseline assessment of all outcomes (T0); (2) A 6-month intervention period, with repeated assessments of all outcomes during the last two weeks of months 3 (T1) and 6 (T2). (3) A 12 month follow up (T3),
  Arms: control

SUMMARY:
Insomnia is a chronic mental health condition characterized by difficulty initiating and maintaining sleep with a prevalence of over 50% in Israeli adults ages 65 and above. It is associated with increased risks for chronic illnesses (e.g., cardiovascular disease), poor mental health (e.g., anxiety and depression), functional limitations, and cognitive decline. Available pharmacological and behavioral treatments focusing on reducing nighttime hyper-arousal offer limited success, and it appears that there is no "one size fits all" treatment for late life insomnia. Mounting evidence suggests that sleep is related to metabolic status, however, studies on the associations between sleep and dietary patterns are surprisingly scarce.

The ability of gut microbiota to communicate with the brain is emerging as an exciting concept in health and disease and provides the rationale for the present project. Findings demonstrate that gut microbiota modulates mental capacities such as brain plasticity and cognitive functions in older adults, as well as stress related mental illness. The composition of the intestinal microbiota in older people (>65 years) differs from the core microbiota and diversity levels of younger adults. With age, gut populations of beneficial microbes show a marked decline. As diet has been shown to markedly promote microbiota biodiversity, it is hypothesized that diet-induced changes in microbiota may provide a novel approach for the treatment of mental health. Although insomnia is strongly linked to mental health (e.g., depression and anxiety), as well as cognitive and motor performance, the effects of diet-induced microbiota alterations, based on individual microbiota composition, on late life insomnia is currently unknown.

The proposed project will be the first to investigate the associations between gut microbiota and sleep, and assess the potential of a six-months personalized, diet-induced microbiota alterations intervention (PDM), aimed to improve insomnia in older adults. We will also look at cognitive, motor and mental health factors as possible mediators in this relationship. Specifically, we will test the associations between microbiota composition and sleep quality, both cross-sectionally and longitudinally, i.e., following a PDM intervention; evaluate the impact of PDM on changes in cognitive, motor and mental health functions; and identify the mediating roles of changes in cognitive, motor and mental functioning on the effects of a PDM intervention on sleep quality. Findings are expected to improve the quality of life of older adults by enhancing their sleep, functional status, mental health and overall wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Based on DSM-5 criteria of diagnosed chronic insomnia in adults, participants will be included if they report difficulties in initiating or maintaining sleep or early morning awakening at least three nights per week that lasts for a minimum of three months, and impaired daytime functioning.

Exclusion Criteria:

* Based on standard clinical history questionnaires and sleep questionnaires, participants will be excluded if they are less than 65 years, have any significant visual or hearing impairments or chronic pain, if they have or had significant and unstable medical, neurological, or psychiatric illness, if they are alcohol or drug abusers or taking psychiatric medication, or if they had sleep apnea syndrome (SAS) or periodic limb movement disorder during sleep (PLMD).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
ISI - Insomnia sevirity Index | one year
  Insomnia Severity Index is based on DSM-4 carteria for insomnia surveys will be completed once at all four study waves (T0-T3)
Actigraphy based Insomnia | one year
  Objective sleep measurements: Actigraphy: wrist-worn ambulatory device/ To obtain a composite score for insomnia based on actigraphy, the following cutoff will be used: sleep efficiency<=85%; and sleep onset latency (SOL) and/or wake after sleep onset (WASO) >=30 minutes, at least 3 times per week.
  Two- week assessments will be repeated during all four study waves (T0-T3)

SECONDARY OUTCOMES:
Insomnia by the consensus sleep diary | one year
  To obtain a composite score for insomnia based on the consensus sleep diary, the following cutoff will be used: sleep efficiency<=85%; and sleep onset latency (SOL) and/or wake after sleep onset (WASO) >=30 minutes, at least 3 times per week.
  Two- week assessments will be repeated during all four study waves (T0-T3)
Insomnia by the The Pittsburgh Sleep Quality Index | one year
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month time interval. Its composite global score is the sum of 7 subscore domains of sleep quality.
  will be completed once at all four study waves (T0-T3)
Cognitive Functioning | one year
  Cognitive performance will be evaluated using the computerized "Cantab connect research" neuropsychological examination for neurocognitive evaluation, which consists of three 20-minute sessions that measure a wide variety of cognitive The Cantab connect research computerized neurocognitive evaluation was specially developed to provide a sensitive test to detect reduction in cognitive functioning among older adults, and it simultaneously provides several measures of cognitive functioning. The software is easy to use and self-explanatory-it guides the user, describes progress rates, and points out areas of difficulty. Assessments will be repeated at all study waves (T0-T3).
Motor Assessment- Gait | one year
  Gait will be evaluated as a composite score based on walking speed and stride variability, as a single task, and together with a cognitive task (e.g., subtraction by 3) as a dual task.
  once at all four study waves (T0-T3)
Motor Assessment- Activity | one year
  Daily activity assessment will be based on a composite score of step count and energy expenditure.
  once at all four study waves (T0-T3)
Wellbeing and Mental health status | one year
  Wellbeing will be assessed using the World Health Organization Quality of Life short form questionnaire (WhoQOL-BREF). These assessments will be carried out at all study waves (T0-T3).
Mental health status - Depression | one year
  Depression will be assessed using the Geriatric Depression Scale (GDS). These assessments will be carried out at all study waves (T0-T3).
Mental health status - Anxiety | one year
  Anxiety will be assessed using the ZUNG selfrating and anxiety scale These assessments will be carried out at all study waves (T0-T3).

OTHER OUTCOMES:
Clinical and nutritional data collection - Anthropometric measures | one year
  Anthropometric measures (height, weight, calf and mid-arm circumference) will be carried out on all participants. Assessments will be repeated at all study waves (T0-T3)
Eating Behavior Questionnaire (CEBQ) | one year
  Appetite, gastrointestinal problems, and chewing and swallowing problems will be assessed using the Composite Eating Behavior Questionnaire (CEBQ). Anthropometric measures (height, weight, calf and mid-arm circumference) will be carried out on all participants. Assessments will be repeated at all study waves (T0-T3)
Nutritional data collection - Food Frequency Questionnaire (FFQ) | one year
  Habitual dietary intake information that will be assessed using the Food Frequency Questionnaire (FFQ). Assessments will be repeated at all study waves (T0-T3)
Microbiota profile | 6 month
  Microbiota composition will be characterized from participants' stools samples collected in the homes. For each assessment, the dietitian will provide the participants with clear guidelines for stools collection,and will collect the specimens during her home visit and immediately put in buffer and store at -80ºC for later usage. The very low temperature is of significance to avoid variability in the stool bacterial composition and to preserve bacterial DNA in fecal samples. Samples will be shipped frozen at -20° to the lab where they will be stored at -80 °C. Total microbial DNA will be extracted using the PowerSoil DNA extraction kit (MoBio) and then submitted to 16S rRNA gene amplicon sequencing. Sequences will be analyzed using the QIIME and MOTHUR pipelines, and data will be integrated into the mega-database.Assessments will be repeated at 3 study waves (T0-T2)

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Shochat, DSc, Principal Investigator — University of Haifa; Uzi Milman, MD, Principal Investigator — Clalit; Iris Haimov, Professor, Principal Investigator — The Max Stern Yezreel Valley College; Maayan Agmon, Ph.D, Principal Investigator — University of Haifa; Snait Tamir, Ph.D, Principal Investigator — Migal, Galilee Technology Center
Locations (1):
- University of Haifa, Haifa, Mount Carmel, Israel

IPD SHARING:
Plan to Share IPD: Undecided